CLINICAL TRIAL: NCT05574088
Title: Comparison of Postoperative Pain With or Without Apical Patency Technique in Asymptomatic Necrotic Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prime Foundation (Other)
Responsible Party: Principal Investigator, Iftikhar Akbar, Professor, Prime Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PrimeF
Record Dates: First submitted 2022-09-16; First posted 2022-10-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; Acute Pain
Keywords: Apical patency; Asymptomatic necrotic teeth,; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Intervention Model Description: !) apical patency 2) Control group ( Non apical patency )
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apical patency (Experimental): 30 patients will be in apical patency group
  Interventions: Procedure: Apical patency with file
- Control group ( non apical patency) (No Intervention): 30 patients will be in control group ( non apical patency)

INTERVENTIONS:
Procedure: Apical patency with file — After an informed consent , One group will receive apical patency intervention with k file number 10 while the other will be control group
  Arms: apical patency

SUMMARY:
Apical patency is a technique in which the apical portion of the canal is maintained free of soft tissue remnants and dentinal debris by recapitulation with a small #10k file through the apical foramen. The purpose of this study is to evaluate the association between apical patency and postoperative pain in teeth with asymptomatic necrotic pulp among patients attending the Peshawar Dental College and Hospital. This single center, double blinded prospective RCT study will be conducted in Peshawar Dental College and Hospital. The inclusion criteria will be mature maxillary and mandibular molars and premolars diagnosed with asymptomatic necrotic pulp and apical periodontitis among 18-60 aged male and female patients, whereas pregnant patients, individuals with previously accessed teeth, and those having positive history of analgesic use within past 3 days will be excluded from the study. A total of 60 patients, after an informed consent will be randomly allocated one of the two groups i.e., apical patency (AP)(n = 30) and the non-apical patency (NAP) (n = 30) in a ratio (1:1).After administering localanaesthesia, root canal preparation will be completed using ProTaper rotary instruments.A size 10 K-filewas carried 1 mm beyond the working length in the patency groupused as a patency file.Patients will be asked to mark their pain intensity on 0-10 scale (NRS)for 7 days. Data will be analyzed using ChiSquare test, Student t-test, Kolmogorov-Smirnov test.

DETAILED DESCRIPTION:
Cleaning and shaping is an integral part of root canal therapy that involves mechanical instrumentation and irrigation of root canal system.1 The apical portion of root canal system is challenging to properly prepare and debride with mechanical instrumentation because of anatomical complexity 2. Dentinal and pulpal debris can be pushed to apical portion during mechanical instrumentation of root canal system, blocking access to apical third which may lead to procedural errors such as loss of working length, perforations, ledge formation and transportation.3, 4 Accumulation of pupal and dentinal debris causing blockage in apical third of the root canal can be prevented only when patency of apical foramen is maintained through apical patency file technique 2, 4, 5.

Apical patency (AP) is a technique in which the apical portion of the canal is maintained free of debris by recapitulation with a small file through the apical foreman 4, 6 thus preventing incidence of procedural accidents, maintaining the required working lengths, improving tactile sensation and facilitating irrigation of apical third of the canal 3-5, 7. In-case of infected or necrotic pulp, it also helps remove the bacterial biofilms around the apical foramen 2, 4. It's importance was also reflected from study conducted by Arias et al there was less postoperative pain when AP was maintained in non-vital pulp 5. Patency file also results in less gas bubbles presented in root canal during cleaning and shaping procedures that could resultin less contact of irrigation solutions with the root canal walls 7, 8.

To maintain apical patency a small flexible K-file (usually a size #10) is set at 1 mm longer than the final working length is intentionally and passively moved through the apical constriction without binding and widening it after each instrument before irrigation.3-5, 9, 10 One of the problems associated with maintaining apical patency is the possible displacement of infected debris through the apical foramen causing acute apical inflammatory response that may lead to postoperative pain2, 5, 9. Furthermore, it may result in damage and transportation of the apical foramen11. However, no such complication as postoperative pain or damage and transportation of apical foramen, resulted 12,13.

Several studies have evaluated the effect of maintaining apical patency on postoperative pain. When patency was maintained in teeth with nonvital pulp, Arias et al5 reported significantly less postoperative pain; however, the author did not describe the periapical status of teeth. While in another RCT did not reveal any significant difference in postoperative pain in teeth with necrotic pulp and apical periodontitis; however, Arora et al13 conducted the study on 68 participants. In addition, the canals preparation was either carried out with hand files 5 or continuous rotary system 13. In a study by Yaylali at al3, who also reported significantly less postoperative pain for first 5 days while maintaining patency; however, the author used reciprocating system for canal preparation and VAS scale for pain severity. In addition, the teeth were not asymptomatic pre-operatively. While in another RCT by Shubham at al18 reported significantly higher pain while maintaining apical patency.

Considering the limitations and conflicting results in previous studies. Hence, this study hypothesizes that there is no difference in terms of post-operative pain between either maintaining apical patency or not. This RCT was designed to evaluate the effect of maintaining apical patency on postoperative pain in teeth with pre-operatively asymptomatic necrotic pulp and apical periodontitis. The primary outcome measure of this study will be to determine the incidence and severity of post-operative pain in both apical patency and non-patency groups; and secondary outcome measure will be to assess post-operative use of analgesics in both groups.

This study will be conducted after the approval from the Institutions of Prime Foundation, a prospective randomized clinical study will be planned at Operative Dentistry and Endodontics Department from 01 Jan, 2021 to 30June, 2021 This single center, double blind prospective RCT study will be conducted in Peshawar Dental College and Hospital. The inclusion criteria will be mature mandibular and maxillary molars and premolars diagnosed with asymptomatic necrotic pulp and apical periodontitis, among 18-65 aged male and female patients.Whereas pregnant patients,complications during treatment (calcified canals, inability to achieve apical patency in any canal), individuals with previously accessed teeth, and those having positive history of analgesic use within past 3 days will be excluded from the study.The pulpal status of each tooth diagnosed as asymptomatic necrotic pulp after clinical examination i-e negative response to cold and electric pulp tests will be confirmed later by absence of bleeding upon endodontic access preparation.

The sample size calculation indicated that a minimum of 30 patients in each group would be sufficient to detect clinically significant differences in pain level, with alpha kept at 0.05,power at 90%, and effect size of 0.8.

After confirming eligibility, the patients will be thoroughly briefed about the study design and the clinical procedure, as well as the associated risks. They will also assured that necessary treatment would be performed regardless of whether they opted to participate in the study or not. Once the patient agreed to participate in the study, written and verbal informed consent will be obtained, and the patients will be randomly allocated one of the two groups i.e., apical patency (AP) and the non-apical patency (NAP) in an equal proportion allocation ratio(1:1) using envelopes that contained sequentially assigned concealed assignment codes to eligible patients. Before access to the root canal system was made, both the patients and the operator will be blinded to the treatment assignment.

The entire root canal procedures will be performed by single operator in all patients. After the root canal procedure,the assessment of post-operative pain will be done through pain scoring chart i.e., the patients will be asked to mark their pain intensity on 0-10 scale and then will be categorised accordingly as no pain (0), mild (1-3), moderate (4-6) and severe (7-10), during 7 days post-operative duration. The pain scale will be thoroughly explained to the patients,and will be given instructions how to use it.The level of pain will be defined as follows:

* mild pain: any discomfort of any duration that does not require the use of analgesics.
* moderate pain: pain that requires analgesics and is only relieved after taking analgesics.
* intense pain: any pain level that is not relieved even after taking the recommended analgesics.

The recommended medication for pain will be ibuprofen(400 mg every 6-8 h). The patients will be given local anaesthesia (2% lidocainewith 1: 100 000 epinephrine) using a conventionalinferior alveolar nerve block.The following standard treatment procedure steps will be followed for all patients. The tooth to be treated will be isolated using rubber dam. Caries removal and access preparation will be carried out using sterile diamond burs with high-speed and air water coolant spray at all times. Root canals will be flared using Low-speed Gates-Glidden burs (Dentsply Maillefer, Ballaigues, Switzerland). Working length will be determined twice during the procedure using electronic apex locator (Root ZX II;J. Morita USA, Inc) with #10 and 15 k-files. The file will be gently advance into the canal until the display on the apex locator indicated 'APEX'. The file will be withdrawn slightly until the display indicated flashing point between 'APEX' and 1. A parallel and angled digital radiographs will be taken to confirm the working length and to verify that the file tip will be within 0.5-1.5 mm of the radiographic apex.The rubber stop on the file will be adjusted to the reference point and the length was measured as working length (WL). Canals will be shaped with ProTaper Universal rotary instruments using finishing files F1, F2, F3 or F4 following the manufacturer'sinstructions. After shaping with finishing file F1, the apical preparation will be assessed with a #20 K-file. The preparation will be deemed to be appropriate,if the file will snug at length. If the file will loose at length, the preparation will be further enlarged with finishing file F2, and even with F3or F4 instruments when deemed necessary after gauging each finishing file with the corresponding hand file until a snug fit at working length will be obtained.

In the patency (AP) group, the patency file, a#10 K-file will be passed 1 mm beyond the WL between each successive instrument used, while in the non-patency (NAP) group it will be carried up to the WL for recapitulation. In the AP group to confirm patency, a final digital radiograph will be taken after completion of preparation,with a #10 K-file placed 1 mm beyond the WL. During the procedure, irrigation will be performed with 5 mL 3% sodium hypochlorite after each instrument using a 30-G endodontic needle (Max-i-Probe, Dentsply Maillefer).After completion of preparation, the canals will be irrigated with 5 mL 17% EDTA for 1 minute followed by 5 ml 3% sodium hypochlorite as a final rinse. The canals will be dried with sterile absorbent paper points, and the canals will be filled with calcium hydroxide paste made by mixing calcium hydroxide powder (Roth International Ltd, Chicago,IL, USA) with distilled water. The tooth will then temporary restored with Cavit W (3 M ESPE, St. Paul, MN, USA).

Patients will be informed of possibility of experiencing pain in the days following treatment and were given instructionto record their pain at 24 h, 2, 3, 4, 5, 6 and 7 days following the treatment, and will be asked to submit at the nextappointment, scheduled after 1 week. They will be advised to use analgesics (ibuprofen 400 mg every6-8 h), if in-case of pain. They will be also instructed to record the details of analgesic in takeon the pain scoring form regarding the number of doses required, timing of the dose and whether it provided adequate pain relief or not (yes/no).

Results of groups AP and NAP related to incidence (yes/no), degree(mild, moderate, severe), and length (days) of post-operative pain will be compared, attending to factors: group of teeth (molars, premolar), or position (upper, lower).Baseline characteristics will also be compared. SPSS 22(SPSS Inc, Chicago, IL) will be used for all statistical analyses. The Student t-test will be used to analyze independent samples. The chi-square test will be used to assess the differences between categoric variables. The comparisons will be considered statistically significant at P < .05.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be mature maxillary and mandibular molars and premolars diagnosed with asymptomatic necrotic pulp and apical periodontitis

Exclusion Criteria:

* whereas pregnant patients, individuals with previously accessed teeth, and those having positive history of analgesic use within past 3 days will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
COMPARISION OF POSTOPERATIVE PAIN WITH OR WITHOUT APICAL PATENCY TECHNQIUE IN ASYMPTOMATIC NECROTIC TEETH | Two months
  postoperative pain in patency and non patency groups will be measured and reported through Numerical rating scale from 0 to 10 for 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Rizwan Qureshi, BDS, FCPS, Study Chair — Peshawar Dental College
Locations (1):
- Peshawar Dental College, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No